CLINICAL TRIAL: NCT03407781
Title: IRDye800CW-BBN PET-NIRF in Lower Grade Glioma
Brief Title: IRDye800CW-BBN PET-NIRF Imaging Guiding Surgery in Patients With Lower Grade Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Deling Li (Other)
Collaborators: Peking Union Medical College Hospital (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Deling Li, Vice Chair of Brain Tumor Ward 2, associate professor, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BTHospital-N-008; ZIAEB000073 (NIH)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Glioma
Keywords: fluorescence guided surgery; dual-modality imaging
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: In the first stage, a small proportion of participants receive preoperative 68Ga-IRDye800-BBN PET/CT and then
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-BBN-IRDye800CW PET/NIRF (Experimental): The patients were injected with 40μg/111-148 Mega-Becquerel (MBq) 68Ga-BBN-IRDye800CW in one dose intravenously and then underwent PET scan 30 min later before the operation and intraoperative 1.0 or 2.0 mg/ml BBN-IRDye800CW injected intravenously for near-infrared (NIR) fluorescent imaging-guided surgery.
  Interventions: Drug: 68Ga-BBN-IRDye800CW

INTERVENTIONS:
Drug: 68Ga-BBN-IRDye800CW — PET/NIR fluorescent imaging-guided surgery
  Other Names: IRDye800CW-BBN

SUMMARY:
This is an open-label positron emission tomography/near infrared (PET/NIRF) study to investigate the imaging navigation performance and evaluation efficacy of dual modality imaging probe 68Ga-BBN-IRDye800CW in patients with lower grade glioma. A single dose of 40μg/111-148 Mega-Becquerel (MBq) 68Ga-NOTA-BBN and 1.0- or 2.0- mg/ml IRDye800CW-BBN will be injected intravenously before the operation and intraoperative respectively. Visual and semiquantitative method will be used to assess the PET images and real-time margins localization for surgical navigation.

DETAILED DESCRIPTION:
Lower grade gliomas (WHO grades II and III) are currently diffused disease with variability of tumor behaviors and of challenge to distinguish the margins in white-light microscope during the surgery. An integrated dual-modality approach combining preoperative positron emission tomography imaging with intraoperative optical guidance that target the same tumor biomarker would be of grade help to solve this problem. BBN, with the amino acid sequence of Gln-Trp-Ala-Val-Gly-His-Leu-Met-NH2, has been extensively used for the development of molecular probes for the imaging of gastrin-releasing peptide receptor (GRPR), a member of the G protein-coupled receptor family of bombesin receptors that over-expressed in various types of cancer cells including glioma. For interests in clinical translation of GRPR targeting dual modality probe, an open label dual modality imaging PET/ NIRF study was designed to investigate the imaging guiding performance in lower grade glioma patients. To investigate whether the preoperative PET with BBN can predict the success of the fluorescence guided surgery with same peptide intraoperatively. The sensitivity, specificity and accuracy of fluorescence guided sampling intraoperatively according to the final pathology will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to provide a written informed consent
* suspected lower grade gliomas on contrast-enhanced MRI

Exclusion Criteria:

* Consisted of conditions of mental illness
* Severe liver or kidney disease with serum creatinine > 3.0 mg/dl (270 μΜ)
* Any hepatic enzyme level 5 times or more than normal upper limit
* Severe allergy or hypersensitivity to IV radiographic contrast
* Claustrophobia to accept the PET/CT or PET/MRI scanning
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-BBN-IRDye800CW in PET imaging of lower grade gliomas | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in lower grade glioma will be measured.

SECONDARY OUTCOMES:
The sensitivity and specificity of intraoperative IRDye800CW-BBN fluorescence | 1 year
  The sensitivity and specificity of intraoperative IRDye800CW-BBN fluorescence, and the preoperative PET and MRI imaging indicator for IRDye800CW-BBN fluorescence imaging in lower grade gliomas

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Study Director — Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College; Nan Ji, MD, Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China